CLINICAL TRIAL: NCT05126082
Title: Improving Recognition and Management of Hypertension in Youth: Comparing Approaches for Extending Effective CDS for Use in a Large Rural Health System
Brief Title: Pediatric Blood Pressure Clinical Decision Support Tool (PedsBP CDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Essentia Health (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EH 20669
Record Dates: First submitted 2021-10-07; First posted 2021-11-18 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: Clinical Decision Support; Hypertension; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: 40 community-based, primary care clinics with the largest number of visits among youth 6-17 years will be balanced and randomly allocated in a 1:1:1 allocation ratio to usual care, low-intensity implementation, or high-intensity implementation of the PedsBP CDS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Providers and patients in control arm clinics will engage in the current standard of care, without access to the PedsBP clinical decision support tool.
- Low-Intensity Implementation (Experimental): Providers and patients in the low-intensity arm will have access to the PedsBP clinical decision support tool and will receive standard training and training resources using the health systems standard training platform.
  Interventions: Behavioral: PedsBP CDS
- High-Intensity Implementation (Experimental): Providers and patients in the high-intensity arm will have access to the PedsBP clinical decision support tool and will receive enhanced training and training resources, and regular feedback from the project team regarding CDS use rates.
  Interventions: Behavioral: PedsBP CDS

INTERVENTIONS:
Behavioral: PedsBP CDS — The PedsBP CDS is a sophisticated web-based electronic health record (EHR)-linked tool that can be used to address barriers and improve the identification and management of elevated blood pressure (BP) and hypertension (HT) in children and adolescents by providing patient-specific clinical care recommendations in real time and in accordance with national guidelines for BP management in youth.
  Arms: High-Intensity Implementation; Low-Intensity Implementation

SUMMARY:
The goal of the PedsBP CDS research project is to adapt a previously tested web-based clinical decision support tool that appropriately identifies high blood pressure in youth for use in a primarily rural health system and compare approaches to CDS implementation in 45 primary care clinics treating children in 3 upper Midwest states. This project will advance implementation science and address a critical need for youth at risk for cardiovascular disease and with limited access to pediatric subspecialty care.

DETAILED DESCRIPTION:
Hypertension (HT) in youth tracks into adulthood, contributing to adult cardiovascular morbidity and mortality. National guidelines for the diagnosis and treatment of HT in children and adolescents were last updated in 2017, with definitions for HT that vary by age. To date, most children and adolescents with elevated blood pressure (BP) or HT are not diagnosed or inadequately treated. Factors that contribute to these deficits in care include: the need to translate pediatric BP measures into BP percentiles, lack of clinician familiarity with pediatric HT guidelines, and competing demands at clinical encounters.

Electronic health record (EHR)-linked clinical decision support (CDS) can be used to address these barriers and improve the identification and management of elevated BP and HT in children and adolescents. In a previous study, the investigators developed, implemented, and evaluated a sophisticated web-based, EHR-linked CDS to provide patient-specific clinical care recommendations in real time and in accordance with national guidelines for BP management in youth. In a 2-year cluster randomized trial in 20 urban and suburban primary care clinics in an integrated health system in Minnesota, the investigators demonstrated that the CDS increased repeat measurement of elevated BP during a visit and more than doubled clinician recognition of HT, while promoting dietitian referrals and additional next steps in care consistent with national guidelines. The CDS system was well accepted by providers and as such, is now standard of care in 55 primary care and 17 subspecialty clinics serving children across our health system. Implementation of this CDS in a new health system is a logical next step, yet optimal strategies for adaptation and implementation of CDS in clinics serving rural populations have not been well described.

In this study, the investigators will implement PedsBP CDS in a large health system with many clinics located in rural regions of Minnesota, Wisconsin and North Dakota. In order to compare approaches to implementation of PedsBP CDS to usual care, the investigators will randomly assign 15 primary care clinics to receive high-intensity implementation (CDS with online and in-person training, and audit-feedback), 15 clinics to receive low-intensity implementation (CDS with online training only), and 15 clinics will continue with usual care (no CDS).

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the PedsBP CDS if

1. 6-17 years of age
2. BP measured and entered in the vital sign section during an ambulatory primary care visit in a randomized primary care clinic
3. not pregnant or postpartum

Patients must meet these eligibility criteria to be included into study analyses:

1. have at least one index visit with a primary care provider at a randomized clinic in the intervention period
2. meet eligibility for PedsBP CDS at index visit (a-c above)
3. no previous HT diagnosis prior to index visit
4. not taking antihypertensive medication prior to index visit
5. not opted out of use of their data for research via general consent prior to performing analyses

Primary care providers must meet these eligibility criteria to participate in this study:

1. practice at a randomized primary care clinic
2. be a pediatric or family medicine care provider (pediatrician, family physician, nurse practitioner or physician assistant), and
3. provide ongoing clinical care for children and adolescents

Exclusion Criteria:

Patients will be excluded from analyses if the following criteria are met:

1. outside of the inclusion age range (<6 years and ≥18 years) at index visit
2. pregnant or postpartum adolescents during study period
3. known HT diagnosis or taking antihypertensive medication at index visit
4. opted out of use of their data for research via general consent prior to performing analyses

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41054 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse O Kharbanda, MD, MPH, Principal Investigator — HealthPartners Institute; Catherine Benziger, MD, MPH, Principal Investigator — Essentia Health
Locations (1):
- Essentia Health, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Providers did not give consent and are not included in the enrollment number. Only patient participants were considered enrolled. Patient participants received care in line with the study arm/group assignment of the primary care clinic in which they received care.
Units Other Than Participants: Primary Care Clinics
Groups:
- Control: Primary care clinics were assigned to control arm clinics and will engage in the current standard of care, without access to the PedsBP clinical decision support tool. Providers at those clinics will provide the usual standard of care.
- Low-Intensity Implementation: Primary care clinics in the low-intensity arm will have access to the PedsBP clinical decision support tool and provider and clinic staff will receive standard training and training resources using the health systems standard training platform.
  PedsBP CDS: The PedsBP CDS is a sophisticated web-based electronic health record (EHR)-linked tool that can be used to address barriers and improve the identification and management of elevated blood pressure (BP) and hypertension (HT) in children and adolescents by providing patient-specific clinical care recommendations in real time and in accordance with national guidelines for BP management in youth.
- High-Intensity Implementation: Primary care clinics in the high-intensity arm will have access to the PedsBP clinical decision support tool and providers and clinic staff will receive enhanced training and training resources, and regular feedback from the project team regarding CDS use rates.
  PedsBP CDS: The PedsBP CDS is a sophisticated web-based electronic health record (EHR)-linked tool that can be used to address barriers and improve the identification and management of elevated blood pressure (BP) and hypertension (HT) in children and adolescents by providing patient-specific clinical care recommendations in real time and in accordance with national guidelines for BP management in youth.
Period: Overall Study
Arm/Group | Control | Low-Intensity Implementation | High-Intensity Implementation
Started | 12072; 13 Primary Care Clinics | 13900; 14 Primary Care Clinics | 15082; 13 Primary Care Clinics
Patients Started | 12072; 13 Primary Care Clinics | 13900; 14 Primary Care Clinics | 15082; 13 Primary Care Clinics
Completed | 12072; 13 Primary Care Clinics | 13900; 14 Primary Care Clinics | 15082; 13 Primary Care Clinics
Not Completed | 0; 0 Primary Care Clinics | 0; 0 Primary Care Clinics | 0; 0 Primary Care Clinics

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected on the providers. We report provider actions at the patient level in the outcomes section.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Low-Intensity Implementation | High-Intensity Implementation | Total
Number analyzed (Participants) | 12072 | 13900 | 15082 | 41054
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (3.5) | 11.7 (3.6) | 11.4 (3.5) | 11.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Unknown Sex:
  Control: 1 Low: 2 High: 2
  Participants
    Sex: number analyzed (Participants) | 12071 | 13898 | 15080 | 41049
    Sex: Female | 5975 | 7061 | 7448 | 20484
    Sex: Male | 6096 | 6837 | 7632 | 20565
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 402 | 333 | 299 | 1034
  Not Hispanic or Latino | 11540 | 13441 | 14576 | 39557
  Unknown or Not Reported | 130 | 126 | 207 | 463
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 380 | 409 | 634 | 1423
  Asian | 125 | 93 | 148 | 366
  Native Hawaiian or Other Pacific Islander | 47 | 50 | 52 | 149
  Black or African American | 779 | 280 | 529 | 1588
  White | 10209 | 12609 | 13056 | 35874
  More than one race | 172 | 157 | 264 | 593
  Unknown or Not Reported | 360 | 302 | 399 | 1061
Region of Enrollment [Number; unit: participants]
  United States | 12072 | 13900 | 15082 | 41054

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Remeasurement
Description: Number of participants with blood pressure re-measurement at the index primary care encounter, among those with a first elevated blood pressure at the index primary care encounter.
Time Frame: Within the index primary care encounter
Population: This is the subset of patients with elevated blood pressure.
Measure: Number; unit: participants
Groups:
- Control: Providers and patients assigned to control arm clinics will engage in the current standard of care, without access to the PedsBP clinical decision support tool.
Arm/Group | Control | Low-Intensity Implementation | High-Intensity Implementation
Number analyzed (Participants) | 3051 | 2903 | 3201
participants | 245 | 829 | 1813
Statistical Analysis 1: Comparison: Control vs Low-Intensity Implementation vs High-Intensity Implementation; Generalized linear mixed models (logit link and binomial error distribution) were used to test the effect of the intervention on blood pressure re-measurement. A planned contrast of the Low + High study arms vs. UC study arm was tested in a model that included pre-specified covariates and a random intercept for clinic. The test of the contrast was 2-sided with p<0.05 considered statistically significant; Test type: Superiority; p < 0.001, Mixed Models Analysis; Denominator degrees of freedom for fixed effects in the model take into account the cluster-randomized design; Adjusted OR = 8.70
Statistical Analysis 2: Comparison: Low-Intensity Implementation vs High-Intensity Implementation; Generalized linear mixed models (logit link and binomial error distribution) were used to test the effect of the intervention on blood pressure re-measurement. A planned contrast of the Low vs High study arms was tested in a model that included pre-specified covariates and a random intercept for clinic. The test of the contrast was 2-sided with p<0.05 considered statistically significant; Test type: Superiority; p < 0.001, Mixed Models Analysis; Denominator degrees of freedom for fixed effects in the model take into account the cluster-randomized design; Adjusted OR = 3.45

2. Primary Outcome: Hypertension Recognition
Description: Number of participants with recognition of hypertension within 6 months of meeting incident hypertension criteria. Clinical recognition of hypertension was based on having a diagnosis of elevated BP (R03) or hypertension (I10, I15) or by having these diagnoses added to the problem list.
Time Frame: Within 6 months of the index primary care encounter at which criteria for incident hypertension were met.
Population: The analytic sample is the subset of patients who newly met criteria for hypertension and had height measured.
Measure: Number; unit: participants
Arm/Group | Control | Low-Intensity Implementation | High-Intensity Implementation
Number analyzed (Participants) | 94 | 186 | 298
participants | 22 | 37 | 121
Statistical Analysis 1: Comparison: Control vs Low-Intensity Implementation vs High-Intensity Implementation; Generalized linear mixed models (logit link and binomial error distribution) were used to test the effect of the intervention on hypertension recognition. A planned contrast of the Low + High study arms vs. UC study arm was tested in a model that included pre-specified covariates and a random intercept for clinic. The test of the contrast was 2-sided with p<0.05 considered statistically significant; Test type: Superiority; p = 0.049, Mixed Models Analysis; Denominator degrees of freedom for fixed effects in the model take into account the cluster-randomized design; Adjusted OR = 2.94
Statistical Analysis 2: Comparison: Low-Intensity Implementation vs High-Intensity Implementation; Generalized linear mixed models (logit link and binomial error distribution) were used to test the effect of the intervention on hypertension recogntion. A planned contrast of the Low vs High study arms was tested in a model that included pre-specified covariates and a random intercept for clinic. The test of the contrast was 2-sided with p<0.05 considered statistically significant; Test type: Superiority; p = 0.03, Mixed Models Analysis; Denominator degrees of freedom for fixed effects in the model take into account the cluster-randomized design; Adjusted OR = 2.31

ADVERSE EVENTS:
Time Frame: Safety events were passively monitored every 6 months during the 18-month intervention period and 12-month follow up period. Patients were monitored for events occurring within 6 months of index visit newly meeting stage 1 and 2 hypertension criteria.
Description: We conducted passive safety surveillance for patients in control and intervention sites using routinely collected electronic health record data to monitor for potential safety events. We did not gather safety information on providers.
  Safety data was gathered on all 596 patients who newly met criteria for hypertension.
Arm/Group | Control | Low-Intensity Implementation | High-Intensity Implementation
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/189 | 0/310
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/189 | 0/310
Other Adverse Events (participants affected / at risk) | 4/97 | 7/189 | 28/310
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=97) | Low-Intensity Implementation (N=189) | High-Intensity Implementation (N=310)
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 0 (0)
Transient Ischemic Attack (Vascular disorders) | 0 (0) | 0 (0) | 0 (0)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=97) | Low-Intensity Implementation (N=189) | High-Intensity Implementation (N=310)
Echocardiogram conducted (Surgical and medical procedures) | 2 (2) | 2 (2) | 8 (8)
Renal Ultrasound Conducted (Surgical and medical procedures) | 0 (0) | 3 (3) | 1 (1)
Hospitalization for any cause (General disorders) | 0 (0) | 1 (1) | 11 (11)
Order for anti-hypertensive medication (Vascular disorders) | 2 (2) | 1 (1) | 8 (8)

LIMITATIONS AND CAVEATS:
The study was conducted in a large, primarily rural health system. Study results may not be generalizable to other health systems, especially those with different structures or urban settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05126082/Prot_SAP_000.pdf